CLINICAL TRIAL: NCT04917094
Title: Effectiveness of Compression Stocking on Overnight Fluid Shift in Obstructive Sleep Apnea Patients
Brief Title: Effectiveness of Compression Stocking on Overnight Fluid Shift in Obstructive Sleep Apnoea Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khoo Teck Puat Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/00393
Record Dates: First submitted 2021-05-31; First posted 2021-06-08 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2022-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Stockings, Compression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Below the knee compression stocking (Experimental)
  Interventions: Device: Compression stocking

INTERVENTIONS:
Device: Compression stocking — A below-the-knee compression stock will be worn daily for 2 weeks from waking up to before sleep.
  Bioelectrical impedance will be performed before and 2 weeks after wearing the stocking to assess the total body water content.
  Measuring the calf and neck circumference will be done before and after wearing the compression stocking. After 2 weeks, the patient will return back to the clinic for calf and neck circumference measurement.
  Sleep test will be done the night before and 2 weeks after wearing the compression stocking. Oxygen Desaturation Index(ODI) will be assessed through a level 4 home sleep apnea testing device.
  Patients recruited will have mild excessive to severe excessive daytime sleepiness and/or STOP-Bang score of 3 or more, with underlying conditions such as type II diabetes and hypertensive patients using the Epworth sleepiness scale. Epworth sleepiness scale will be assessed again 2 weeks after to assess for increase sleep efficiency.

SUMMARY:
Overnight rostral fluid shift is one of the contributing factors for worsening obstructive sleep apnoea (OSA). Fluid shift has been recognized to play a role in the pathophysiology of sleep apnoea. Previous studies shown that fluid from the leg redistributes to the neck at night increases the neck circumference, hence indicating fluid accumulation in the neck. OSA patients are more susceptible to developing upper airway narrowing in response to fluid shift from the leg to the head and neck region.

Previous studies were mainly done on Caucasian patients. The pathophysiology of OSA in Caucasian patients and Asian patients are different but both suffer a similar degree of OSA. The investigators would like to investigate if reducing leg swelling by a simple non-invasive intervention of wearing compression stocking during the day can attenuate sleep apnoea, and whether compression stocking is generally acceptable and well-tolerated among the general OSA population in Asia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 years old to 65 years old.
* Either STOP-Bang score of ≥3 or Epworth sleepiness scale indicating mild excessive daytime sleepiness to severe excessive daytime sleepiness (11-24 points).
* Has pre-existing diabetes mellitus and/or hypertension and is on medication.
* Ability to provide informed consent.
* Not working night shift.

Exclusion Criteria:

* Significant arterial disease due to the risk of limb ischaemia and necrosis.
* Not pregnant and not planning to get pregnant before the end of the study.
* History of psychiatric disease.
* Patient who are on wheelchair.
* Patient who has cardiac failure and or stroke.
* Patient who has end-stage renal failure. Estimated glomerular filtration rate <15ml/min/1.73m2 or on renal replacement therapy i.e. dialysis or renal transplant.
* Patient who has liver disease.
* Patient who are on pacemaker, and metal implants.
* Patient who are on CPAP treatment for OSA.
* Patient who are illiterate.
* Medications which affect fluid balance or level of consciousness (e.g. diuretics, non- steroidal anti-inflammatory drugs (NSAIDS), corticosteroids, sedatives, opiates) at any time during the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Compression stocking improves ODI of OSA patients | 2 weeks
  Bioelectrical impedance analysis (BIA) readings performed before wearing the compression stocking and 2 weeks after wearing the compression stocking to assess the total body water, lower limb total water content (LLW), lower limbs extracellular water content (ecLLW), trunk total water content (TW), trunk extracellular water content (ecTW), neck fluid volume and leg fluid volume will be improved.
  Calf and neck circumference measurements before wearing the compression stocking and 2 weeks after wearing the compression stocking will be improved.
  Sleep test done to measure the Oxygen Desaturation Index (ODI) the night before wearing the compression stocking and 2 weeks before the final visit to the clinic will be improved.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Seet, Principal Investigator — Khoo Teck Puat Hospital
Locations (1):
- Khoo Teck Puat Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Friedman O, Bradley TD, Chan CT, Parkes R, Logan AG. Relationship between overnight rostral fluid shift and obstructive sleep apnea in drug-resistant hypertension. Hypertension. 2010 Dec;56(6):1077-82. doi: 10.1161/HYPERTENSIONAHA.110.154427. Epub 2010 Nov 8. PMID 21060007
- [Result] Gonzaga C, Bertolami A, Bertolami M, Amodeo C, Calhoun D. Obstructive sleep apnea, hypertension and cardiovascular diseases. J Hum Hypertens. 2015 Dec;29(12):705-12. doi: 10.1038/jhh.2015.15. Epub 2015 Mar 12. PMID 25761667
- [Result] Perger E, Jutant EM, Redolfi S. Targeting volume overload and overnight rostral fluid shift: A new perspective to treat sleep apnea. Sleep Med Rev. 2018 Dec;42:160-170. doi: 10.1016/j.smrv.2018.07.008. Epub 2018 Aug 4. PMID 30177246
- [Result] Reutrakul S, Mokhlesi B. Obstructive Sleep Apnea and Diabetes: A State of the Art Review. Chest. 2017 Nov;152(5):1070-1086. doi: 10.1016/j.chest.2017.05.009. Epub 2017 May 17. PMID 28527878
- [Result] da Silva BC, Kasai T, Coelho FM, Zatz R, Elias RM. Fluid Redistribution in Sleep Apnea: Therapeutic Implications in Edematous States. Front Med (Lausanne). 2018 Jan 22;4:256. doi: 10.3389/fmed.2017.00256. eCollection 2017. PMID 29404327
- [Result] White LH, Lyons OD, Yadollahi A, Ryan CM, Bradley TD. Night-to-night variability in obstructive sleep apnea severity: relationship to overnight rostral fluid shift. J Clin Sleep Med. 2015 Jan 15;11(2):149-56. doi: 10.5664/jcsm.4462. PMID 25406274
- [Result] White LH, Lyons OD, Yadollahi A, Ryan CM, Bradley TD. Effect of below-the-knee compression stockings on severity of obstructive sleep apnea. Sleep Med. 2015 Feb;16(2):258-64. doi: 10.1016/j.sleep.2014.12.005. Epub 2014 Dec 18. PMID 25620198
- [Result] White LH, Bradley TD. Role of nocturnal rostral fluid shift in the pathogenesis of obstructive and central sleep apnoea. J Physiol. 2013 Mar 1;591(5):1179-93. doi: 10.1113/jphysiol.2012.245159. Epub 2012 Dec 10. PMID 23230237
- [Result] Redolfi S, Arnulf I, Pottier M, Bradley TD, Similowski T. Effects of venous compression of the legs on overnight rostral fluid shift and obstructive sleep apnea. Respir Physiol Neurobiol. 2011 Mar 15;175(3):390-3. doi: 10.1016/j.resp.2011.01.001. Epub 2011 Jan 8. PMID 21220055
- [Result] Redolfi S, Arnulf I, Pottier M, Lajou J, Koskas I, Bradley TD, Similowski T. Attenuation of obstructive sleep apnea by compression stockings in subjects with venous insufficiency. Am J Respir Crit Care Med. 2011 Nov 1;184(9):1062-6. doi: 10.1164/rccm.201102-0350OC. PMID 21836140
- See also: Impact of Compression Stockings vs. Continuous Positive Airway Pressure on Overnight Fluid Shift and Obstructive Sleep Apnea among Patients on Hemodialysis — https://www.frontiersin.org/articles/10.3389/fmed.2017.00057/full
- See also: Night-to-night Variability in Obstructive Sleep Apnea Severity: Relationship to Overnight Rostral Fluid Shift — https://doi.org/10.5664/jcsm.4462